CLINICAL TRIAL: NCT02341209
Title: Doxycycline in Patients With Relapsed Cutaneous T-cell Lymphoma
Brief Title: Doxycycline for the Treatment of Cutaneous T-Cell Lymphoma
Acronym: CTCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, Brian Poligone, MD, PhD, Scientist II, Rochester General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53677
Record Dates: First submitted 2014-11-21; First posted 2015-01-19 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cutaneous T-cell Lymphoma; Mycosis Fungoides; Sezary Syndrome
Keywords: CTCL; Sezary Syndrome (SS); Mycosis Fungoides (MF); Cutaneous T-cell Lymphoma; MF; SS
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Doxycycline

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doxycycline monohydrate (Experimental): Doxycycline in either capsules or tablets will be administered at 400mg total per day. Patients will be treated for five months, or up to one year for those with a partial response at 5 months.
  Interventions: Drug: Doxycycline monohydrate

INTERVENTIONS:
Drug: Doxycycline monohydrate — Doxycycline will be administered in either tablets or capsules for either five months or a year depending on response.
  Other Names: Adoxa, Mondox

SUMMARY:
This study looks at the efficacy of Doxycycline for the treatment of Cutaneous T-cell Lymphomas.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of doxycycline in relapsed Cutaneous T-cell Lymphomas (CTCL). The primary objective is to determine the overall response rate of doxycycline monotherapy in patients with relapsed CTCL.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated Institutional Review Board approved informed consent form in accordance with regulatory and institutional guidelines. Written informed consent must be obtained prior to performing any study-related procedure.
* Be 18 years of age or older at time of enrollment.
* Measurable disease in at least one target lesion in the skin or able to be assessed by radiographic examination with FDG-PET fluorodeoxyglucose possitron emission tomography (FDG-PET) scan or computarized tomography (CT) scan, or peripheral blood showing involvement of lymphoma.
* The subject has resolution of all clinically significant toxic effects of prior cancer therapy to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI-CTCAE, v.4.0) excluding the specification below.
* Adequate organ function:
* Absolute Neutrophil Count (ANC) > 500 cells/mL and platelet count > 50,000 cells/mL unless felt to be secondary to lymphoma at which any count is permissible.
* Adequate renal function as determined by creatinine < 1.5x upper limit normal (ULN) or estimated creatinine clearance of ≥ 60ml/min
* Adequate hepatic function as determined by total bilirubin < 1.5x ULN (unless known Gilbert syndrome), Alanine transaminase (ALT) and Aspartate transaminase (AST) < 2.5x ULN
* Confirmed diagnosis of CTCL.
* Karnofsky Performance Status ≥ 60%
* Women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days of receiving study medication and monthly while on receiving doxycycline
* WOCBP must agree to use effective contraception, defined as, oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide) or practice true abstinence from sexual intercourse (periodic abstinence, e.g., calendar ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception) during the study and for 3 months after the last dose. WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea ≥ 12 consecutive months without an alternative medical cause).
* Male subjects and their female partners of child bearing potential must be willing to use an appropriate method of contraception defined as, oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide) or practice true abstinence from sexual intercourse (periodic abstinence, e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception) during the study and for 3 months after the last dose.

Exclusion Criteria:

* Known sensitivity or allergy to tetracyclines
* Lack of measurable disease
* Karnofsky Performance Status <60%
* Inadequate organ function as measured by not fulfilling above criteria
* Subject is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Doxycycline in relapsed CTCL | From baseline to five month or a year depending on response.
  Overall response rate will be determined after five months or a year from initiation of therapy.

SECONDARY OUTCOMES:
Duration of Response | From baseline to up to one year.
  Patients who achieve a Partial Response or Complete Response will be monitored for progression up to one year after initiation of therapy.

OTHER OUTCOMES:
Quality of Life evaluation | Baseline to up to one year.
  Changes in quality of life will be measured throughout the study using questionnaires.
Pruritus (Itchiness) evaluation | Baseline to up to one year.
  Changes in quality of life will be measured throughout the study using questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Poligone, M.D. Ph.D., Principal Investigator — Rochester General Hospital
Locations (1):
- Rochester General Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
As required